CLINICAL TRIAL: NCT07392541
Title: A Single-Arm, Multicenter, Exploratory Clinical Study of Adebrelimab in Combination With Gemcitabine, Cisplatin, and Simvastatin for the Treatment of Patients With Locally Advanced or Metastatic Biliary Tract Malignancies
Brief Title: Adebrelimab Combined With Gemcitabine, Cisplatin, and Simvastatin for Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-07
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Carcinoma
Keywords: Advanced Biliary Tract Carcinoma; adebrelimab; simvastatin
MeSH Terms: interventions — Gemcitabine; Cisplatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Intervention (Experimental): All participants receive the combination therapy of adebrelimab, gemcitabine, cisplatin, and simvastatin for up to 8 cycles (21-day/cycle), followed by maintenance therapy with adebrelimab and simvastatin until disease progression or unacceptable toxicity.
  Interventions: Drug: Adebrelimab; Drug: Gemcitabine + Cisplatin; Drug: Simvastatin 20mg

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab is an anti-PD-L1 monoclonal antibody. During the initial combination phase (up to 8 cycles), it is administered intravenously at 1200 mg on Day 1 of each 21-day cycle. During the subsequent maintenance phase, it is administered at 1200 mg intravenously every 4 weeks.
  Other Names: SHR-1316
Drug: Gemcitabine + Cisplatin — Standard gemcitabine and cisplatin chemotherapy regimen. This combination is administered intravenously only during the initial treatment phase for a maximum of 8 cycles (21-day cycles).
  Other Names: GemCis
Drug: Simvastatin 20mg — Simvastatin is an HMG-CoA reductase inhibitor (statin). It is administered orally at a dose of 20 mg once daily continuously throughout both the initial combination phase and the subsequent maintenance phase until treatment completion criteria are met.

SUMMARY:
This study will investigate the safety and effectiveness of a new combination treatment for patients with advanced bile duct cancer. The treatment combines standard chemotherapy drugs (gemcitabine and cisplatin) with two additional medications: adebrelimab and simvastatin.

All participants in this study will receive the same four-drug combination. Researchers will closely monitor patients to see how well the tumors shrink, how long the treatment keeps the cancer from growing, and what side effects occur. The study is exploratory, meaning it aims to gather initial data on whether this four-drug combination is a promising approach for treating advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed unresectable, locally advanced, or metastatic biliary tract adenocarcinoma (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer).
* No prior systemic therapy for advanced disease if initially diagnosed as unresectable or metastatic. Disease recurrence occurring more than 6 months after radical surgery or adjuvant therapy is allowed.
* ECOG Performance Status of 0 or 1.
* At least one radiologically measurable lesion as defined by RECIST 1.1 criteria (tumor lesion with longest diameter ≥10 mm on CT scan, or lymph node with short axis ≥15 mm).
* No severe dysfunction of major organs (heart, lungs, brain, etc.).

Exclusion Criteria:

* Diagnosis of ampullary carcinoma.
* Presence of active or previously documented autoimmune or inflammatory disorders.
* Known hypersensitivity to any component of the study drugs (adebrelimab, gemcitabine, cisplatin, simvastatin).
* Severe liver dysfunction: laboratory tests within 14 days prior to enrollment showing total bilirubin > 1.5 times the upper limit of normal (ULN), AND/OR alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times ULN.
* Participation in another investigational drug or device clinical trial within 4 weeks prior to enrollment.
* Inability to comply with the study protocol for treatment or scheduled follow-up assessments.
* Any other condition deemed by the investigator as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment until the first documented disease progression or completion of study treatment, whichever occurs first, assessed up to approximately 2 years.
  The proportion of participants achieving a best overall response of Complete Response (CR) or Partial Response (PR) according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Tumor assessments will be performed by investigators via contrast-enhanced CT or MRI scans.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment until the first documented progression or death from any cause, assessed up to approximately 2 years
  PFS is defined as the time from the start of study treatment to the first documented disease progression according to RECIST 1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | From enrollment until death from any cause, assessed up to approximately 3 years.
  OS is defined as the time from the start of study treatment to death from any cause.
Disease Control Rate (DCR) | From enrollment until the first documented disease progression or completion of study treatment, assessed up to approximately 2 years.
  DCR is defined as the proportion of participants achieving a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (lasting for at least 6 weeks) according to RECIST 1.1.
Duration of Response (DOR) | From the first documented response until disease progression or death, assessed up to approximately 2 years.
  DOR is defined as the time from the first documentation of objective response (CR or PR) to the first documented disease progression or death from any cause, whichever occurs first, in participants who achieve a confirmed response.
Incidence of Treatment-Related Adverse Events (TRAEs) | From the first dose of study treatment until 30 days after the last dose, assessed up to approximately 2 years.
  The proportion of participants experiencing any adverse event determined by the investigator to be related to the study treatment regimen. Severity is graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No